CLINICAL TRIAL: NCT01061190
Title: Beta-Blocker in Acute Ischemic Stroke - a Prospective, Randomized, Double-blinded, Placebo-controlled Safety and Efficacy Trial of Early Treatment
Brief Title: Beta Blockers In Acute Ischemic Stroke
Acronym: BIAS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wilhelm Haverkamp (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Wilhelm Haverkamp, MD, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BIAS1.0; ZS EK 11 165/09 (Other: ethic's committee of the German federal state Berlin); 2008-007031-41 (EudraCT Number)
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Active Comparator)
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator)
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — oral application of 160 mg Propranolol for 30 days

SUMMARY:
The objective of this trial is to assess the safety and efficacy of neuro- and cardioprotective effects of propranolol in acute ischemic stroke. Furthermore, exploratory analyses of cardiologic-electrophysiologic and immunologic parameters will be performed.

DETAILED DESCRIPTION:
The main objective of this trial is to assess the efficacy and safety of propranolol in middle cerebral artery stroke patients. The primary hypothesis is as follows: Early administration of propranolol reduces the frequency of cardiovascular and/or neurological complications including vascular death in the first 30 days after acute ischemic stroke. Secondary hypotheses are as follows: Early administration of propranolol improves neurological and functional outcome of patients with acute ischemic stroke. Early administration of propranolol reduces post-stroke immunodepression and therefore lowers the rate of pneumonia after acute ischemic stroke, without increasing the frequency of auto-aggressive, CNS antigen-specific T cells. Early administration of propranolol influences alterations in cardiologic, electrophysiologic phenomenons as a reaction to autonomic dysregulation after acute ischemic stroke. Early administration of Propranolol reduces growth of infarct as determined by MRI examinations in the first 6 days.

ELIGIBILITY:
Inclusion Criteria:

* Symptom onset within 18 hours
* Acute ischemic MCA-territory stroke
* Patients with suspected stroke in MCA-territory and a) NIHSS > 3 or b) imaging evidence of MCA-infarction

Exclusion Criteria:

* Patients already receiving beta-blockers
* Anti-arrhythmic, antiinfectious, antiinflammatory or immunosuppressive therapy
* Patients with a major heart disease, hypotension, bradycardia or any contraindication to the use of Propranolol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
composite incidence of cardiovascular and/or neurological complications including vascular death | 90 days

SECONDARY OUTCOMES:
mRS and lethality | 90 days
number of SAEs and treatment withdrawals | 90 days
immunological & cardiological parameters | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Haverkamp, Prof. Dr. med., Principal Investigator — Charité, University Berlin, Center for Stroke Research Berlin
Locations (1):
- Charité, University Berlin, Center for Stroke Research Berlin, Berlin, State of Berlin, Germany